CLINICAL TRIAL: NCT07081945
Title: Prospective Study on the Use of Human Amniotic Membrane (hAM) in the Treatment of Inferior Rhegmatogenous Retinal Detachment (RRD)
Brief Title: hAM for Inferior RRD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hAM for inferior RRD
Record Dates: First submitted 2025-07-22; First posted 2025-07-24 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Rhegmatogenous Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hAM (Experimental): This is a single arm study using literature-reported postoperative outcomes of IRB-RRD patients as the comparator.
  Interventions: Device: hAM

INTERVENTIONS:
Device: hAM — The hAM stands for human amniotic membrane, which was used to seal inferior retinal breaks after complete vitrectomy.

SUMMARY:
The objective of the study is to evaluate the efficacy of using hAM patches over the retina to seal inferior retinal breaks. The researchers will evaluate whether hAM patch-assisted vitrectomy improves surgical success rate of retinal reattachment.

DETAILED DESCRIPTION:
Rhegmatogenous retinal detachments (RRDs) with inferior retinal breaks (IRB-RRD) still remains a challenge with relatively high risk of primary surgical failure and recurrent RRDs. Actually, the single-operation success rate for inferior RRD ranges from 60 % to 90 % as reported. Human amniotic membrane (hAM) and has been reported to be safe for intraocular use, such as macular hole and ocular open globe injury.

Researchers previously reported a 'sandwich' technique for flattening and positioning large-sized hAM patches over the retina, which allowed surgeons to select the optimal hAM size intraoperatively based on surgical need, and thus expanding the application of hAM in RRD. Researchers had demonstrated that covering the exposed retinal pigment epithelium (RPE) with a large-size hAM graft effectively prevented postoperative proliferative vitreoretinopathy (PVR) by the 'sandwich' technique.

This study will include 50 patients with IRB-RRD, who will be treated with hAM patch-assisted vitrectomy, in which hAM patches will be used to seal inferior retinal breaks over the retina after complete vitrectomy. Then researchers will conduct no less than 6 months follow-up and evaluate whether hAM patch-assisted vitrectomy improves surgical success rate of retinal reattachment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects having given free and informed consent to take part in the study.
2. Subjects between 18 and 70 years old.
3. Subjects suffering RRD (both primary and recurrent RRDs) with at least one of these conditions:

   1. inferior retinal breaks between 4- and 8-o'clock within the detached area regardless of PVR grade;
   2. requiring retinotomy inferiorly between 4- and 8-o'clock (due to severe inferior PVR or inferior retinal shortening).

Exclusion Criteria:

1. Subjects with RRD with only anterior retina breaks or dialysis and meet the indications for scleral buckling surgery.
2. Subjects with RRD whose retinal breaks located between the 4- and 8-o'clock positions and are not involved in the detached area.
3. Subjects with pre-existing serious eye diseases (corneal ulcers, glaucoma, uveitis, etc).
4. History of epilepsy or serious psychiatric diseases.
5. Other conditions that the researcher found improper to be included into this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Retinal reattachment rate | From enrollment to the end of the 6-month follow-up period.
  The percentage of patients who achieved retinal reattachment after undergoing hAM patch-assisted vitrectomy during the 6-month follow-up period.
Visual acuity improvement | From enrollment to the end of the 6-month follow-up period.
  The visual acuity improvement 6 months after the surgical procedure measured by Snellen chart.

CONTACTS AND LOCATIONS:
Locations (1):
- EyeEntFudan, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Utra-wide fundus image data of patients pre and postoperatively may be shared with other researchers.
Supporting Information: Study Protocol
Time Frame: After start of recruiting patients.